CLINICAL TRIAL: NCT05610111
Title: Adaptive Biobehavioral Control (ABC) in a Closed-Loop System: A Randomized Crossover Clinical Trial
Brief Title: Adaptive Biobehavioral Control (ABC) in a Closed-Loop System
Acronym: ABC-WIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sue Brown (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Sue Brown, Study Physician, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 220300; 2R01DK085623 (NIH)
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Closed-Loop Control (CLC); Continuous Glucose Monitoring (CGM); Artificial Pancreas (AP); Tandem t:slim Insulin Pump with Control-IQ Technology
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- CLC, then CLC+BAM, then CLC+ABC (Active Comparator): Participants will be using closed loop control (CLC) for 2 weeks. Participants will then use closed loop control (CLC) with behavioral adaption module (BAM) for 4 weeks, followed by closed loop control (CLC) adaptive biobehavioral control (ABC) for 16 weeks.
  Interventions: Device: CLC + BAM; Device: CLC + ABC
- CLC+ABC, then CLC+BAM, then CLC (Active Comparator): Participants will be using closed loop control (CLC) with adaptive biobehavioral control (ABC) for 16 weeks. Participants will then use closed loop control (CLC) with behavioral adaptation module (BAM) for 4 weeks, followed by closed loop control (CLC) for 2 weeks.
  Interventions: Device: CLC + BAM; Device: CLC + ABC

INTERVENTIONS:
Device: CLC + BAM — Closed Loop Control with the Behavioral Adaption Module for 4 weeks
Device: CLC + ABC — Closed Loop Control with Adaptive Biobehavioral Control for 16 weeks

SUMMARY:
This study is intended to test a Web-based Information Tool (WIT) software providing additional information regarding time in range, GMI, hypo- and hyperglycemia risks, variability tracker, daily glycemic profiles, and potential changes of insulin pump parameters, to users of a commercially available Closed-Loop Control (CLC) System (Control-IQ Technology).

DETAILED DESCRIPTION:
This is a randomized two-arm crossover group trial in which both groups will use the CLC (Control-IQ) plus WIT. The difference between the two groups will be the order of the interventions. Each group will undergo screening and collection of baseline data from their personal AID system (Control-IQ) followed by randomization 1:1 into two groups. Both groups will have the same three interventions but will progress in the study in a different order allowing for crossover comparisons. The three interventions are:

* Use of personal CLC system for 2 weeks
* Use of personal CLC system and adding a behavioral adaptation module (BAM) for 4 weeks
* Use of personal CLC system and adding the ABC which includes: BAM and PAM (which includes ATM and WST described below) for 16 weeks.

The BAM will consist of modules in which information only is given to participants (e.g. time in range, Glucose Management Indicator (GMI), hyper-and hypoglycemic risks, daily glycemic profiles, and variability tracker). The PAM includes auto suggestions for titration of insulin pump parameters every two weeks (ATM) and is aided by a web simulation tool (WST) which can replay 'what if' scenarios for the participant based on various combinations of insulin pump parameter changes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.0 and ≤70 years old at time of consent
2. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year
3. Currently using an insulin pump for at least six months
4. Currently using insulin for at least six months
5. Currently using the t:slim X2 insulin pump for at least two months
6. Currently using or anticipated to be using the t:slim X2 insulin pump with Control-IQ technology at randomization (Visit 3).
7. Using or willing to use insulin parameters such as carbohydrate ratio and correction factors consistently on their pump in order to dose insulin for meals or corrections
8. Access to internet and willingness to upload data during the study as needed
9. Willing to use an app on a smart phone during the study.
10. For females, not currently known to be pregnant or breastfeeding
11. If female, sexually active, and of childbearing potential, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of childbearing potential. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
12. Willingness to use only insulin analogs approved for use in the t:slim X2 pump such as lispro (Humalog) or as part (Novolog) and not use ultra-rapid acting insulin analogs (e.g., FiAsp) during the study
13. Total daily insulin dose (TDD) at least 10 units per day
14. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial (including metformin (biguanides), GLP-1 receptor agonists, pramlintide, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas)
15. An understanding and willingness to follow the protocol and signed informed consent

Exclusion Criteria:

1. Concurrent use of any non-insulin glucose-lowering agent other than metformin or GLP-1 receptor agonists following screening (including pramlintide, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas)
2. A condition, which in the opinion of the investigator or designee, would put the participant at risk or interfere with the completion of the protocol.
3. History of diabetic ketoacidosis (DKA) in the 12 months prior to enrollment
4. Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment
5. Currently being treated for a seizure disorder
6. Hemophilia or any other bleeding disorder
7. Planned surgery during study duration
8. Participation in another pharmaceutical or device trial at the time of enrollment or during the study
9. Having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (e.g., study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
CGM-measured percent time in range 70-180 mg/dL | 4 weeks
  The primary outcome for this study is CGM-measured percent time in range 70-180 mg/dL over the last 4-week periods on CLC+ABC versus 2 weeks of the current CLC system. The intervention will be considered effective if the CLC+ABC is superior to the CLC alone in a crossover design using a statistical significance of α=0.05.
  To preserve the overall type 1 error for selected key secondary endpoints, a hierarchical testing procedure will be used. If the primary analysis for time in range described above results in a statistically significant result (p < 0.05), then testing (similar to the model for the primary outcome) will proceed to the next key secondary outcome metric in the following order entered.

SECONDARY OUTCOMES:
CGM-measured percent above 180 mg/dL during the day | 4 weeks
  A key secondary outcome is CGM-measured percent above 180mg/dL during the day comparing last 4 weeks of CLC+ABC to 2 weeks of the CLC system alone. If the analysis results in a statistically significant result (p < 0.05), then testing will proceed to the next secondary outcome metric in the following order entered.
CGM-measured percent below 70 mg/dL during the day | 4 weeks
  A key secondary outcome is CGM-measured percent below 70 mg/dL during the day comparing last 4 weeks of CLC+ABC to 2 weeks of the CLC system alone. If the analysis results in a statistically significant result (p < 0.05), then testing will proceed to the next secondary outcome metric in the following order entered.
CGM-measured mean glucose | 4 weeks
  A key secondary outcome is CGM-measured mean glucose comparing the last 4 weeks of CLC+ABC to 2 weeks of the CLC system alone. If the analysis results in a statistically significant result (p < 0.05), then testing will proceed to the next secondary outcome metric in the following order entered.
CGM-measured coefficient of variation during the day | 4 weeks
  A key secondary outcome is CGM-measured percent coefficient of variation during the day comparing last 4 weeks of CLC+ABC to 2 weeks of the CLC system alone.

CONTACTS AND LOCATIONS:
Overall Officials: Sue Brown, MD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance. Limited deidentified data will be shared while sharing of complete data sets will be regulated by Data-Sharing Agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Generally following completion of publications.
Access Criteria: Limited deidentified data will be shared while sharing of complete data sets will be regulated by Data-Sharing Agreements.

REFERENCES:
- [Result] Kovatchev BP, Colmegna P, Pavan J, Diaz Castaneda JL, Villa-Tamayo MF, Koravi CLK, Santini G, Alix C, Stumpf M, Brown SA. Human-machine co-adaptation to automated insulin delivery: a randomised clinical trial using digital twin technology. NPJ Digit Med. 2025 May 6;8(1):253. doi: 10.1038/s41746-025-01679-y. PMID 40329052

DOCUMENTS (1):
  • Informed Consent Form (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT05610111/ICF_000.pdf